CLINICAL TRIAL: NCT06795893
Title: Pregnancy and Infant Outcomes in Anifrolumab Exposed Pregnancies Using PRegnancy Outcomes Intensive Monitoring (PRIM) Data: The Anifrolumab PRIM Program
Brief Title: The Anifrolumab PRIM Program
Acronym: PRIM
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00090
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: chronic autoimmune disease; immunosuppressants; corticosteroids; human monoclonal antibody (IgG1ƙ mAb); post Marketing Requirements (PMR) study; pregnancy; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anifrolumab exposed pregnancies: The primary analysis cohort will be prospectively reported pregnancies with anifrolumab exposure anytime from 16 weeks prior to date of conception (DOC) until pregnancy outcome.
  Interventions: Drug: Anifrolumab

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab is a human monoclonal antibody that binds to subunit 1 of the type 1 interferon receptor,which was developed based on the evidence supporting the role of type 1 interferon pathway in SLE. Clinical trial evidence from TULIP 1 and TULIP 2 have showed that monthly intravenous administration of anifrolumab led to a higher percentage of patients with a response, assessed with the British Isles Lupus Assessment Group-based Composite Lupus Assessment, compared with patients receiving placebo. Moreover, the phase II MUSE study showed that administration of anifrolumab resulted in substantially reduce disease activity, as measured by the SLE Responder Index,compared to patients receiving placebo. Anifrolumab was approved by the FDA and EMA in July 2021 and February 2022,respectively, for the treatment of adult patients with moderate to severe SLE who are receiving standard therapy.
  Other Names: Saphnelo

SUMMARY:
Pregnancy and infant outcomes in anifrolumab exposed pregnancies using PRegnancy outcomes Intensive Monitoring (PRIM) data: The anifrolumab PRIM program

DETAILED DESCRIPTION:
The anifrolumab PRIM program is a supplementary program which utilizes enhanced collection of secondary data from reported anifrolumab-exposed pregnancies collected as part of AstraZeneca's PV system.

Initial information about the exposed pregnancy will be collected through the pregnancy report submitted by anifrolumab treated patients or HCPs to the AstraZeneca PV database. Pregnancy outcome information will be collected in close proximity to the planned delivery. Additional follow-up and outcome information will be collected 12 months after delivery. For PV reports of exposed pregnancies that have already had a pregnancy outcome at the time of initial report (retrospective cases), initial characteristics, pregnancy outcome, and any available infant health information will be collected at the time of the initial report.

Targeted follow-up checklists and guidance documents will ensure that PV data collected for anifrolumab-exposed pregnancies are as complete as possible and have been mapped for pre-specified analytic variables that will be used to evaluate the safety of anifrolumab exposure for pregnancy and infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently or recently (within 1 year of pregnancy outcome) pregnant
* Exposure to at least 1 dose of anifrolumab at any time during pregnancy or in the 16 weeks prior to date of conception

Exclusion Criteria:

* Pregnancy cases that have been enrolled in the prospective pregnancy registry (D3461R00051), those reported prior to the start of the PRIM program, or those that have been exposed to known teratogens or investigational medications will be excluded from the anifrolumab PRIM study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pregnancies exposed to anifrolumab and reported to the AstraZeneca pharmacovigilance database on or after the initiation of the PRIM program, regardless of when the pregnancy outcome was ascertained.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2031-04-15 (Estimated); Study Completion 2031-04-15 (Estimated)

PRIMARY OUTCOMES:
Major congenital malfunctions | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  The primary objective of the PRIM program is to estimate the proportion of anifrolumab-exposed pregnancies with major congenital malformations (MCMs) associated with exposure to anifrolumab during pregnancy.

SECONDARY OUTCOMES:
Minor congenital malformations | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  To estimate the proportion of anifrolumab-exposed pregnancies with minor congenital malformations associated with exposure to anifrolumab during pregnancy.
Adverse pregnancy outcomes | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  To estimate the proportion of anifrolumab-exposed pregnancies with adverse pregnancy outcomes and adverse birth outcomes associated with exposure to anifrolumab during pregnancy.
Frequency of adverse pregnancy and birth outcomes | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  To estimate the frequency of adverse pregnancy and birth outcomes associated with exposure to anifrolumab during pregnancy and adverse effects on immune system development in infants with follow-up of up to one year of age.

CONTACTS AND LOCATIONS:
Overall Officials: Syd Philips, Principal Investigator — PPD Miami, US
Locations (1):
- Reseach Facility, Södertälje, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/